CLINICAL TRIAL: NCT01070420
Title: Comparison of Hyperemic Efficacy Between Central and Peripheral Adenosine Infusion for Fractional Flow Reserve (FFR) Measurement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Bon- Kwon Koo / prof, Cardiovascular Center, Seoul National University Hospital,
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: D-0910-002-062
Record Dates: First submitted 2010-01-10; First posted 2010-02-18 (Estimated); Last update posted 2011-07-18 (Estimated); Status verified 2011-07

CONDITIONS: Coronary Artery Disease; Myocardial Ischemia
Keywords: Adenosine; Fractional flow reserve, Hyperemia; Fractional Flow Reserve, Myocardial
MeSH Terms: conditions — Coronary Artery Disease; Myocardial Ischemia; Hyperemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- FFR via central venous line (Active Comparator)
  Interventions: Other: FFR via central venous line
- FFR via peripheral vein (Experimental)
  Interventions: Other: FFR via peripheral venous line

INTERVENTIONS:
Other: FFR via central venous line — Patients with intermediate coronary artery stenosis were consecutively enrolled. FFR was measured by a standard intravenous (IV) adenosine infusion (140 μg•min-1•kg-1) via Rt central femoral vein.
  Arms: FFR via central venous line
Other: FFR via peripheral venous line — Patients with intermediate coronary artery stenosis were consecutively enrolled. FFR was measured by a standard intravenous (IV) adenosine infusion (140 μg•min-1•kg-1) via continuous peripheral vein.
  Arms: FFR via peripheral vein

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of the peripheral IV continuous infusion without the insertion of central venous vascular access method in the achievement of steady-state maximal coronary hyperemia compared with the central IV continuous infusion method.

ELIGIBILITY:
Inclusion Criteria:

* non -infarct related, patients with moderate coronary artery stenosis
* normal ejection fraction on echocardiogram

Exclusion Criteria:

* infarct-related arteries or clinically unstable state
* collateral blood flow to the target vessel is shown
* atrioventricular block on electrocardiogram
* reduced ejection fraction(<50%) or left ventricular hypertrophy on echocardiography
* contraindication of adenosine

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2009-12; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
compare fractional flow reserve at maximal hyperemia | interval of 10 minutes

SECONDARY OUTCOMES:
compare the time to maximal hyperemia and changes in heart rate | interval of 10 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Bon- Kwon Koo, MD, PhD, Study Chair — Department of Internal Medicine, Cardiovascular Center, Seoul National University Hospital
Locations (1):
- Cardiovascular Center, Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Park DW, Kim YH, Song HG, Ahn JM, Kim WJ, Lee JY, Kang SJ, Lee SW, Lee CW, Park SW, Yun SC, Her SH, Hur SH, Park JS, Kim MK, Choi YS, Kim HS, Cho JH, Lee SG, Park YW, Jeong MH, Lee BK, Lee NH, Lim DS, Yoon J, Seung KB, Shin WY, Rha SW, Kim KS, Tahk SJ, Park BE, Ahn T, Yang JY, Jeong YS, Rhew JH, Park SJ; IRIS-DES Investigators. Outcomes after unrestricted use of everolimus-eluting and sirolimus-eluting stents in routine clinical practice: a multicenter, prospective cohort study. Circ Cardiovasc Interv. 2012 Jun;5(3):365-71. doi: 10.1161/CIRCINTERVENTIONS.111.966549. Epub 2012 Jun 12. PMID 22693347
- [Derived] Seo MK, Koo BK, Kim JH, Shin DH, Yang HM, Park KW, Lee HY, Kang HJ, Kim HS, Oh BH, Park YB. Comparison of hyperemic efficacy between central and peripheral venous adenosine infusion for fractional flow reserve measurement. Circ Cardiovasc Interv. 2012 Jun;5(3):401-5. doi: 10.1161/CIRCINTERVENTIONS.111.965392. Epub 2012 May 29. PMID 22647519